CLINICAL TRIAL: NCT06080347
Title: An Evaluator-blinded Randomized Controlled Trial Study of the Effect of Anti-inflammatory Diet in Subjects With Osteoarthritis
Brief Title: Effect of Anti-inflammatory Diet in Osteoarthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Monica Guma, Associate Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 807845
Record Dates: First submitted 2023-10-06; First posted 2023-10-12 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Diet, Healthy

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm_1 (Active Comparator): Anti-inflammatory Diet
  Interventions: Other: Anti-inflammatory Diet
- Arm_2 (Experimental): Healthy Diet
  Interventions: Other: Healthy Diet

INTERVENTIONS:
Other: Anti-inflammatory Diet — Dietary intervention
  Arms: Arm_1
Other: Healthy Diet — Dietary intervention
  Arms: Arm_2

SUMMARY:
In a previous exploratory study, the investigators observed an effect on disease activity outcomes of anti-inflammatory diet. The investigators also observed change in microbiome and circulating metabolites. The current study will determine whether or not the addition of anti-inflammatory diet improves the clinical outcomes in participants with Osteoarthritis, and the role of microbiome and circulating metabolites.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral radiographic symptomatic KOA
* No changes in therapy during the previous 3 months
* Interested in dietary intervention and able to provide consent and attend follow-up visits

Exclusion Criteria:

* Previous knee surgery
* Severe radiographic disease (KL grade 4)
* Rheumatoid Arthritis
* Any Abnormal blood values in the comprehensive metabolic panel test at screen (Abnormality will be defined based on standard reference ranges)
* Use of corticosteroids and/or intra-articular injections during the preceding 3 months
* Use of fish oils and glucosamine
* Participation in a weight loss program in the preceding 6 months
* Recent changes in physical activity levels
* Regular smoking
* Patients with food allergies
* Patient with other medical conditions that will impair the ability to participate in a nutritional study
* Plan to change systemic therapy
* Patients unwilling to change dietary habits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in Knee Osteoarthritis Pain | 3 months
  The Western Ontario and McMaster Universities Osteoarthritis Index, known as the WOMAC score, is a validated questionnaire used for evaluating pain, stiffness, and physical function in individuals with knee or hip osteoarthritis. A minimum score of 0 indicates no symptoms and a maximum score of 100, represents the most severe symptoms. Higher WOMAC scores correspond to worse outcomes, indicating more significant pain, stiffness, and functional limitations associated with osteoarthritis. The primary outcome for the purpose of this study will be the proportion of patients experiencing a change of at least 30% in WOMAC-pain score after 3 months of intervention compared to the control group.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No